CLINICAL TRIAL: NCT06829979
Title: A Pilot, Feasibility Study to Improve Night Shift Nurses' Health and Reduce Burnout
Brief Title: Improving Night Shift Nurses' Health and Reducing Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Shadyside Hospital Foundation (Other)
Responsible Party: Principal Investigator, Christopher Imes, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY24090069
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: Sleep; Fatigue; Burnout; Night shift
MeSH Terms: conditions — Fatigue; Burnout, Psychological | interventions — RID

STUDY DESIGN:
Intervention Model Description: All participants are in a single group/cohort. Everyone will receive the same interventions in the same order. The order of the interventions will be randomly selected from six possible choices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group, crossover - order of the interventions to be randomly selected (Experimental): All participants will receive the same interventions which includes access to the napping/relaxation room only intervention, blue and green light blocking glasses only intervention, and the combined intervention. There will be a two-week washout between the interventions. The order of the interventions will be randomized to one of the following options:
  * Napping/relaxation room, blue and green light blocking glasses, combined
  * Blue and green light blocking glasses, napping/relaxation room, combined
  * Napping/relaxation room, combined, blue and green light blocking glasses
  * Blue and green light blocking glasses, combined, napping/relaxation room
  * Combined, napping/relaxation room, blue and green light blocking glasses
  * Combined, blue and green light blocking glasses, napping/relaxation room
  Interventions: Behavioral: Access to napping/relaxation room; Other: Blue and green light blocking glasses

INTERVENTIONS:
Behavioral: Access to napping/relaxation room — During the night shift, study participants will have access to the hospital unit's napping/relaxation room with a sound machine, diffusers for aromatherapy, a massage chair that can be used for napping, and snacks.
Other: Blue and green light blocking glasses — During the night shift, participants will be asked wear study-provided blue and green light blocking glasses.

SUMMARY:
Healthy and happy nurses are essential to ensuring optimal patient outcomes and organizational success. The evidence on the negative impacts of night shift on nurses' health and cognitive function, and their implications on patient outcomes and organizational costs, reflect the need for interventions to mitigate these detrimental outcomes.

This pilot, feasibility, clinical trial will examine the feasibility of two fatigue countermeasure interventions (access to napping/relaxation room and use of blue/green light blocking glass during night shift) and explore the interventions effects on nurses' health, missed care, and burnout.

DETAILED DESCRIPTION:
Aim 1 (Primary): Examine the feasibility of a larger study and hospital-wide implementation of two fatigue countermeasure interventions (access to napping/relaxation rooms and use of blue/green light blocking glass during night shift).

Aim 2 (Exploratory): Explore the effects of the interventions on melatonin levels, overall health, sleep, fatigue, cognitive function, missed care, nurse burnout, and salivary melatonin levels.

ELIGIBILITY:
Inclusion Criteria:

* Being a registered nurse at UPMC Shadyside (Pittsburgh, PA)
* Working full-time night or rotating shifts
* Willing to wear a Fitbit around-the-clock during the study
* Willing to use nap/relaxation room and glasses only when assigned to that condition
* Willing to provide saliva samples

Exclusion Criteria:

* Having a diagnosed sleep disorder (e.g., obstructive sleep apnea, insomnia, restless leg syndrome, or shift work disorder)
* Currently being treated for a serious mental illness
* Needing to use eye glasses to complete work related activities (note: contact lenses are acceptable)
* Use of prescription or over-the-counter sleep aides including melatonin

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 2 months
  Number of potential participants screened in order to enroll 8 participants
Attrition rate | 4 months
  Percentage of enrolled participants completing the intervention as a whole and its three conditions
Completeness of questionnaire responses | 4 months
  Percentage of completed responses
Melatonin collection | 4 months
  Number of salivary melatonin samples collected

SECONDARY OUTCOMES:
Changes in physical health between baseline and the three conditions | 3 months
  Changes the in PROMIS Global Health 10-item Measure, Physical Health sub-scale T-score.
  T-score ranges from 16.2 to 67.7 with 50.0 (standard deviation of 10) being the population mean.
  Higher scores represent better physical health.
Changes in mental health between baseline and the three conditions | 3 months
  Changes the in PROMIS Global Health 10-item Measure, Mental Health sub-scale T-score.
  T-score ranges from 21.2 to 67.6 with 50.0 (standard deviation of 10) being the population mean.
  Higher scores represent better mental health.
Changes in Multidimensional Sleep Health between baseline and the three conditions | 3 months
  Changes in RSATED survey scores Total score ranges from 0 to 12 with higher scores representing better sleep health.
Changes in sleep distrubance between baseline and the three conditions | 3 months
  Changes in PROMIS Sleep Disturbance 8-item Measure T-scores. T-score ranges from 28.9 to 76.5.7 with 50.0 (standard deviation of 10) being the population mean.
  Higher scores represent more sleep disturbances.
Changes in sleep-related impairment between baseline and the three conditions | 3 months
  Changes in PROMIS Sleep-related Impairment 8-item Measure T-scores. T-score ranges from 30.2 to 80.1 with 50.0 (standard deviation of 10) being the population mean. Higher scores represent more sleep-related impairment.
Change in sleep duration between baseline and the three conditions | 3 months
  Change in mean actigraphic sleep duration
Change in sleep efficiency between baseline and the three conditions | 3 months
  Change in mean actigraphic sleep efficiency
Change in fatigue between baseline and the three conditions | 3 months
  Change in PROMIS Fatigue 7-item Measure T-scores. T-score ranges from 29.4 to 83.2 with 50.0 (standard deviation of 10) being the population mean. Higher scores represent more fatigue.
Change in cognition function between baseline and the three conditions | 3 months
  Change in PROMIS Cognitive Function 8-item Measure T-scores. T-score ranges from 22.41 to 83.2 with 63.48 (standard deviation of 10) being the population mean. Higher scores represent better cognitive function.
Change in burnout between baseline and the three conditions | 3 months
  Change in Copenhagen Burnout Inventory scores. The Copenhagen Burnout Inventory has three sub-scales measuring personal burnout, work-related burnout, and client-related burnout. Sub-scales scores range from 0 to 100 with higher scores representing greater burnout.
Changes in missed care between baseline and the three conditions | 3 months
  Changes in Tasks Undone-12 Scale scores. Scores range from 0 to 12 with higher scores representing more undone nursing tasks.
Changes in salivary melatonin levels between baseline and the three conditions | 3 months
  Changes in salivary melatonin levels

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Shadyside, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets from the research may be shared.
Access Criteria: A Limited Dataset (LDS) may be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.